CLINICAL TRIAL: NCT02276716
Title: The Nutritional Supplement Phosphatidylserine in Patients With Familial
Brief Title: The Nutritional Supplement Phosphatidylserine in Patients With Familial Dysautonomia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-02100
Record Dates: First submitted 2014-10-16; First posted 2014-10-28 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Familial Dysautonomia
MeSH Terms: conditions — Dysautonomia, Familial | interventions — Phosphatidylserines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Phosphatidylserine (Experimental): Phosphatidylserine titration from 300, 600 and 800 mg/day
  duration: 6 months
  Interventions: Dietary Supplement: Phosphatidylserine

INTERVENTIONS:
Dietary Supplement: Phosphatidylserine — Phosphatidylserine will be titrated starting at 300mg/day dose for two months to 600mg/day dose for 2 months, then 800 mg/day dose for a final 2 month period.

SUMMARY:
Familial dysautonomia (FD) is a devastating hereditary disease in which the development of selective neuronal populations is impaired because of a deficiency of the protein IKAP (Slaugenhaupt, 2002). There is no known cure. Treatments are supportive, often ineffective and around half of all patients die before reaching age 40 (Axelrod et al., 2002).

Phosphatidylserine is an FDA approved food supplement that was shown recently to correct the genetic abnormality and restore IKAP protein levels in cell lines derived from patients with FD (Keren et al., 2011) and a humanized mouse model of the disease (Bochner et al., 2013). Despite its safety and efficacy in this fragile population being unknown, many patients with FD are currently taking phosphatidylserine

The investigators propose to conduct a safety, tolerability and early proof of concept efficacy study of phosphatidylserine in patients with FD. The study will be divided into two independent arms. The first phase of the study will be an open-label dose titration study to determine the safety and optimal dose of phosphatidylserine and its effect of normal IKBKAP mRNA levels in 40 patients with FD. The second phase will be a longitudinal observational study in which we will follow, on a yearly basis, patients with FD of all ages who opt to take phosphatidylserine. In this study, we will evaluate the long-term safety of phosphatidylserine in patients with FD and hope to determine whether phosphatidylserine has any impact on the clinical evolution of the disorder.

Our long-term goal is to find an effective therapy that will improve the quality of life for patients with FD and alter disease prognosis. We believe that the promise of phosphatidylserine and its availability in health food shops warrants a controlled safety, tolerability and efficacy study to determine whether it should be taken by patients with FD. This study is not intended to determine whether phosphatidylserine has a new indication to treat FD.

DETAILED DESCRIPTION:
Familial dysautonomia (FD) is an autosomal recessive disease caused by mutations in the I-B kinase complex associated protein (IKBKAP) gene sequence (Anderson et al., 2001; Slaugenhaupt et al., 2001). The disorder affects the development of sensory nerves, resulting in impaired pain and temperature perception (Riley et al., 1949), lack of visceral sensations (Norcliffe-Kaufmann et al., 2010), dysphagia and proprioceptive gait ataxia (Macefield et al., 2011). Childhood mortality is increased, with aspiration pneumonia a leading cause of death. In early adulthood, renal failure is common (Pearson et al., 1980) and eyesight deteriorates due to optic atrophy and gait ataxia worsens making walking impossible without assistance. The incidence of seizures, scoliosis, respiratory insufficiency, sleep apnea and gastrointestinal bleeds are all increased. Sudden unexpected cardiac deaths are common and there is an increased incidence of cancer. Current treatments are supportive and frequently ineffective. FD has no known cure and 50% of patients die before age 40.

A decade ago, we discovered that the disease was caused by point mutations in IKBKAP gene, leading to a deficiency of I-B kinase complex associated protein (IKAP) mainly in neuronal tissue (Slaugenhaupt et al., 2001; Mezey et al., 2003; Lee et al., 2009). Phosphatidylserine, an FDA-approved food supplement, was shown to increase protein levels in FD-derived cell lines (Keren et al., 2011) as well as in a mouse model of FD (Bochner et al., 2013). Because of the severity of FD, the availability of phosphatidylserine in health food stores and its promise as a treatment, many patients with FD are already taking it, although its safety and efficacy in this population is unknown. Thus, we propose a controlled study of phosphatidylserine to determine its safety profile and whether it has any impact on the natural history of FD.

SPECIFIC AIM 1: It is not known if phosphatidylserine increases the levels of IKBKAP mRNA in patients with FD. To determine the optimal dose of phosphatidylserine in patients with FD, (i.e., the lowest dosage at which there is maximal improvement in IKBKAP mRNA production without significant side effects) we will monitor the safety and efficacy of phosphatidylserine in an open-label dose escalation study. Safety parameters and IKBKAP mRNA levels in blood will be measured in 40 patients with FD at baseline and repeated at increasing doses of phosphatidylserine.

SPECIFIC AIM 2: In an independent long-term observational study, we will follow patients with FD of all ages who opt to take phosphatidylserine as a food supplement in their diet. Safety parameters will be measured as part of routine evaluations on an annual basis. The long-term efficacy of phosphatidylserine will be determined by evaluating the evolution of standard parameters of neurological function overtime in patients who received phosphatidylserine and comparing their progression with historical controls from the database archives.

ELIGIBILITY:
Inclusion Criteria:

* - Diagnosis of familial dysautonomia (with mutation testing)
* Age 12 years or older
* Signed informed consent (or ascent), which will include permission to assess medical records

Exclusion Criteria:

* Patients with significant cardiac, respiratory, or renal compromise that, in the investigators opinion, may jeopardize their health by participating in this trial
* Patients who are currently participating in other clinical trials of compounds that my change IKAP gene expression.
* Women who are pregnant or lactating
* Women of childbearing potential who are not using medically accepted methods of contraception.
* Patients taking anticoagulants, such as warfarin, heparin, aspirin, pentoxifylline, clopidogrel or ticlopidine.
* Patients taking ginko, garlic or vitamin E supplements.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-11; Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in blood lab values at every 2 month interval | measurements will be taken at baseline and at two months intervals for the first 6 months, then at yearly intervals for up to 5 years
  blood lab values, CBC, metabolic panel,physical exam, vital signs, 12 lead ECG
Change from baseline in adverse events measures at every 2 month interval | measurements will be taken at baseline and at two months intervals for the first 6 months, then at yearly intervals for up to 5 years
  number of participants with adverse events
Change from baseline in physical exam measures at every 2 month interval | measurements will be taken at baseline and at two months intervals for the first 6 months, then at yearly intervals for up to 5 years
  change from baseline in physical exam
Change from baseline in 12 lead ECG measures at every 2 month interval | measurements will be taken at baseline and at two months intervals for the first 6 months, then at yearly intervals for up to 5 years
  change from baseline in 12 lead ECG
Change from baseline in vital signs measures at every 2 month interval | measurements will be taken at baseline and at two months intervals for the first 6 months, then at yearly intervals for up to 5 years
  change from baseline in sitting blood pressure, body temperature

SECONDARY OUTCOMES:
Change from baseline in efficacy measures | measurements will be taken at baseline and at two months intervals for the first 6 months, then at yearly intervals for up to 5 years
  Change from baseline in IKBKP mRNA blood levels at each 2 month intervals

CONTACTS AND LOCATIONS:
Overall Officials: Horacio Kaufmann, MD, Principal Investigator — NYU School of Medicine
Locations (1):
- NYU Langone Medical Center, Dyautonomia Center, Suite 9Q, New York, New York, United States